CLINICAL TRIAL: NCT02389088
Title: Effect of Increased Circulating Androgens on Granulosa Cell Responses to FSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Professor Emeritus of Reproductive Medicine Division of Reproductive Endocrinology and Infertility, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UCSD-2016
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Granulosa Cell; Androgens; FSH; Ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (No Intervention): 9 PCOS women will be studied. On study day one, r-FSH will be administered I.V. at a dose of 150 IU (FSH stimulation test). Blood samples will be obtained before and after FSH administration. After the FSH stimulation test, each subject will receive an I.M. injection of Lupron 3.75 mg. This dose has a duration effect of one month.
  The FSH stimulation test will be repeated, as described above, at 5 weeks (early resumption of ovarian function) and 6 weeks (moderate resumption of ovarian function).
- Phase II (Active Comparator): Women that participated in Phase I will be studied again after a washout of 2 months. On study day one, an FSH stimulation test will be performed as described above.
  After the FSH stimulation test, each subject will receive an I.M. injection of Lupron 3.75 mg. This dose has a duration effect of one month. Four weeks after administration of Lupron, each subject will receive Letrozole 5mg for 14 days. The FSH stimulation test will be repeated at 5 weeks (early resumption of ovarian function) and 6 weeks (moderate resumption of ovarian function).
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — In Phase II, letrozole, 5 mg/day, will be given for 14 days
  Other Names: Femora
  Arms: Phase II

SUMMARY:
The purpose of this study is to evaluate the effect of increased circulating androgens on estradiol production by the granulosa cells in response to FSH stimulus.

DETAILED DESCRIPTION:
Various previous studies have demonstrated that androgens enhance granulosa cell function in a variety of animal species including rodents and non-human primates. In vitro studies have shown that granulosa cells exposed to either testosterone or dihydrotestosterone exhibit increased production of estrogen, progesterone and inhibin in response to FSH. Studies done in non-human primates have also shown that androgen increases the numbers of preantral and antral follicles as well as increases FSH receptor mRNA expression in granulosa cells. This suggests that granulosa cell hyperresponsiveness to FSH in polycystic ovary syndrome (PCOS) may be related to androgen excess. The investigators plan to address this possibility by performing a series of in vivo studies. In one of the investigator's prior studies androgen blockade was done by administration of flutamide and E2 responses to FSH assessed. This study has been completed and the manuscript is being prepared for publication. In the present protocol, the investigators propose to further study the role of androgens with a 2 phase study. In the first phase the investigators plan to suppress endogenous steroid hormone production by the ovaries via treatment with the GnRH analog Lupron for 4 weeks beyond which a gradual resumption of ovarian activity will occur. Granulosa cell (inhibin B) responses to FSH will be examined before and after ovarian suppression as well as during early and moderate recovery of ovarian steroidogenesis. These results will provide control data to which comparisons can be made from results of the next phase.

In the second phase, after a 2 month washout interval, the same subjects will again receive Lupron to suppress endogenous steroid production. After 4 weeks, at the beginning of ovarian activity resumption, the investigators will administer Letrozole 5mg for 14 days and again examine granulosa cell responses to FSH during recovery. Letrozole is a 3rd generation aromatase inhibitor which results in suppression of E2 production and increase in circulating serum androgen levels to about 40% greater than pre-treatment values. It is now also being used for ovulation induction. It has minimal side effects and is in general very well tolerated. By using Letrozole for 2 weeks after GnRH suppression of the ovaries, the investigators will more effectively increase the amount of circulating androgen while keeping estrogen at low levels, thereby allowing the investigators to more completely study the effects of isolated and elevated androgen levels on granulosa cell responses to FSH. By comparing results obtained in phase 1, the investigators will be able to determine if there is an androgen mediated response by granulosa cells to FSH stimulation in the absence of other ovarian steroids. Also, the addition of a control group will allow investigators to determine if the granulosa cell response is different between PCOS and normals.

It is hypothesized that there will be a significant rise in inhibin B production by the granulosa cells in PCOS women in response to FSH after treatment with Letrozole as compared to both the control group and to responses observed in the control phase of study. This would confirm that androgens are indeed responsible at least in part for the hyperresponsiveness to FSH seen in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be determined to have PCOS based on clinical criteria such as history of irregular menses and clinical or laboratory evidence of hyperandrogenism.
* Subjects should not have been on any hormonal therapy or metformin for at least 2 months prior to study start.

Exclusion Criteria:

* Women with hemoglobin less than 11gm/dl at screening evaluation.
* Women with untreated thyroid abnormalities
* Pregnant women
* Women with BMI>37
* Women with known sensitivity to the agent being used.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2006-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Jeffrey Chang, M.D., Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Homer MV, Rosencrantz MA, Shayya RF, Chang RJ. The effect of estradiol on granulosa cell responses to FSH in women with polycystic ovary syndrome. Reprod Biol Endocrinol. 2017 Feb 10;15(1):13. doi: 10.1186/s12958-017-0230-0. PMID 28187771

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - All Study Participants: 9 PCOS women will be studied. On study day one, r-FSH will be administered I.V. at a dose of 150 IU (FSH stimulation test). Blood samples will be obtained before and after FSH administration. After the FSH stimulation test, each subject will receive an I.M. injection of Lupron 3.75 mg. This dose has a duration effect of one month.
  The FSH stimulation test will be repeated, as described above, at 5 weeks (early resumption of ovarian function) and 6 weeks (moderate resumption of ovarian function).
Period: Overall Study - Phase I
Arm/Group | Phase I - All Study Participants
Started | 9
Completed | 9
Not Completed | 0
Period: Phase II - All Study Participants
Arm/Group | Phase I - All Study Participants
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 9 PCOS women
Groups:
- Phase I: 9 PCOS women
Arm/Group | Phase I
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — San Diego
  participants
    United States | 9
Phase I - LH, FSH [Mean (Standard Deviation); unit: IU/L]
  LH | 9.5 (4.04)
  FSH | 5.1 (1.03)
Phase I - Testosterone, Androstenedione, 17-OH Progesterone [Mean (Standard Deviation); unit: nmol/L]
  Testosterone | 1.34 (0.3)
  Androstenedione | 5.29 (1.3)
  17-OH Progesterone | 47.3 (24.6)
Phase I - Estradiol [Mean (Standard Deviation); unit: pmol/L] | 180.4 (25.5)
Phase II - LH, FSH [Mean (Standard Deviation); unit: IU/L]
  LH | 8.6 (4.4)
  FSH | 4.7 (1.3)
Phase II - Testosterone, Androstenedione, 17-OH Progesterone [Mean (Standard Deviation); unit: nmol/L]
  Testosterone | 1.3 (0.4)
  Androstenedione | 5.5 (1.6)
  17-OH Progesterone | 53.3 (43.7)
Phase II - Estradiol [Mean (Standard Deviation); unit: pmol/L] | 195.7 (97.4)

OUTCOME MEASURES:

1. Primary Outcome: Estradiol During Phase I and Phase II
Description: Estradiol (pmol/L) measured during Phase I (without Letrozole) and during Phase II (with Letrozole) at time 24 hours during Week 0 and times 0 and 24 hours during Weeks 5 and 6 after FSH stimulation.
Time Frame: At time 24 hours during Week 0 and times 0 and 24 hours during Weeks 5 and 6 after FSH stimulation for both Phase I and Phase II
Population: Phase I and Phase II - PCOS patients.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Phase I - Week 0 - 24 Hours | Phase I - Week 5 - 0 Hour | Phase I - Week 5 - 24 Hour | Phase I - Week 6 - 0 Hour | Phase I - Week 6 - 24 Hour | Phase II - Week 0 - 24 Hours | Phase II - Week 5 - 0 Hours | Phase II - Week 5 - 24 Hours | Phase II - Week 6 - 0 Hours | Phase II - Week 6 - 24 Hours
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
pmol/L | 451.7 (131) | 116 (27.8) | 247.2 (105.5) | 131.4 (20.2) | 347.5 (83.9) | 401.4 (103.4) | 57.9 (27) | 91.3 (80.8) | 66.5 (36.6) | 126.6 (117.7)

2. Primary Outcome: Inhibin B During Phase I and Phase II
Description: Inhibin B (ng/L) measured during Phase I (without Letrozole) and during Phase II (with Letrozole) at time 24 hours during Week 0 and times 0 and 24 hours during Weeks 5 and 6 after FSH stimulation.
Time Frame: as for outcome 1
Population: Phase I and Phase II - PCOS patients.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Phase I - Week 0 - 24 Hours | Phase I - Week 5 - 0 Hour | Phase I - Week 5 - 24 Hour | Phase I - Week 6 - 0 Hour | Phase I - Week 6 - 24 Hour | Phase II - Week 0 - 24 Hours | Phase II - Week 5 - 0 Hours | Phase II - Week 5 - 24 Hours | Phase II - Week 6 - 0 Hours | Phase II - Week 6 - 24 Hours
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
ng/L | 420.6 (120) | 87.9 (76.5) | 395.1 (186.5) | 85.2 (40.2) | 445.5 (169) | 390 (142.4) | 165.2 (202.7) | 340 (309) | 184.3 (192.1) | 427.3 (260)

3. Primary Outcome: LH and FSH During Phase I and Phase II
Description: LH and FSH (IU/L) measured during Phase I (without Letrozole) and during Phase II (with Letrozole) at time 24 hours during Week 0 and times 0 and 24 hours during Weeks 5 and 6 after FSH stimulation.
Time Frame: as for outcome 1
Population: Phase I and Phase II - PCOS patients.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Phase I - Week 0 - 24 Hours | Phase I - Week 5 - 0 Hour | Phase I - Week 5 - 24 Hour | Phase I - Week 6 - 0 Hour | Phase I - Week 6 - 24 Hour | Phase II - Week 0 - 24 Hours | Phase II - Week 5 - 0 Hours | Phase II - Week 5 - 24 Hours | Phase II - Week 6 - 0 Hours | Phase II - Week 6 - 24 Hours
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
IU/L
  LH | NA (NA) — Stimulated value not measured. | 0.6 (0.8) | NA (NA) — Stimulated value not measured. | 2.0 (2.0) | NA (NA) — Stimulated value not measured. | NA (NA) — Stimulated value not measured. | 1.22 (1.8) | NA (NA) — Stimulated value not measured. | 3.6 (3.9) | NA (NA) — Stimulated value not measured.
  FSH | NA (NA) — Stimulated value not measured. | 3.5 (1.2) | NA (NA) — Stimulated value not measured. | 4.3 (0.9) | NA (NA) — Stimulated value not measured. | NA (NA) — Stimulated value not measured. | 8.0 (2.6) | NA (NA) — Stimulated value not measured. | 9.3 (3.1) | NA (NA) — Stimulated value not measured.

4. Primary Outcome: Testosterone, Androstenedione and 17-OH Progesterone During Phase I and Phase II
Description: Testosterone, Androstenedione and 17-OH Progesterone (nmol/L) measured during Phase I (without Letrozole) and during Phase II (with Letrozole) at time 24 hours during Week 0 and times 0 and 24 hours during Weeks 5 and 6 after FSH stimulation.
Time Frame: as for outcome 1
Population: Phase I and Phase II - PCOS patients.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Phase I - Week 0 - 24 Hours | Phase I - Week 5 - 0 Hour | Phase I - Week 5 - 24 Hour | Phase I - Week 6 - 0 Hour | Phase I - Week 6 - 24 Hour | Phase II - Week 0 - 24 Hours | Phase II - Week 5 - 0 Hours | Phase II - Week 5 - 24 Hours | Phase II - Week 6 - 0 Hours | Phase II - Week 6 - 24 Hours
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
nmol/L
  Testosterone | NA (NA) — Stimulated values not measured | 0.6 (0.2) | NA (NA) — Stimulated values not measured | 0.8 (0.4) | NA (NA) — Stimulated values not measured | NA (NA) — Stimulated values not measured | 0.6 (0.2) | NA (NA) — Stimulated values not measured | 0.01 (0.44) | NA (NA) — Stimulated values not measured
  Androstenedione | NA (NA) — Stimulated values not measured | 2.8 (0.9) | NA (NA) — Stimulated values not measured | 3.6 (1.0) | NA (NA) — Stimulated values not measured | NA (NA) — Stimulated values not measured | 2.9 (0.8) | NA (NA) — Stimulated values not measured | 4.3 (1.9) | NA (NA) — Stimulated values not measured
  17OH-Progesterone | NA (NA) — Stimulated values not measured | 32.1 (17.5) | NA (NA) — Stimulated values not measured | 31.1 (9.8) | NA (NA) — Stimulated values not measured | NA (NA) — Stimulated values not measured | 24.0 (16.1) | NA (NA) — Stimulated values not measured | 37.4 (22.1) | NA (NA) — Stimulated values not measured

ADVERSE EVENTS:
Groups:
- Phase II: Women that participated in Phase I will be studied again after a washout of 2 months. On study day one, an FSH stimulation test will be performed as described above.
  After the FSH stimulation test, each subject will receive an I.M. injection of Lupron 3.75 mg. This dose has a duration effect of one month. Four weeks after administration of Lupron, each subject will receive Letrozole 5mg for 14 days. The FSH stimulation test will be repeated at 5 weeks (early resumption of ovarian function) and 6 weeks (moderate resumption of ovarian function).
  Letrozole: In Phase II, letrozole, 5 mg/day, will be given for 14 days
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes